CLINICAL TRIAL: NCT06697938
Title: Neoadjuvant Chemoradiotherapy Compared to Neoadjuvant Chemotherapy for Luminal-Type Locally Advanced Breast Cancer: a Clinical Study
Acronym: NCRT-LABC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sichuan Cancer Hospital and Research Institute (Other)
Responsible Party: Principal Investigator, Qian Peng, Director of the Department of Abdominal Radiotherapy, Ward 1, Sichuan Cancer Hospital and Research Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SCCSMC-01-2024-034
Record Dates: First submitted 2024-11-18; First posted 2024-11-20 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Breast Cancer
Keywords: locally advanced breast cancer; neoadjuvant radiotherapy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Neoadjuvant Chemoradiotherapy Group (Experimental): Preoperative umor SBRT and surgery after Neoadjuvant Chemotherapy
  Interventions: Radiation: Preoperative SBRT for the Primary Lesion of Breast Cancer
- Neoadjuvant Chemotherapy Group (No Intervention): Surgery after Neoadjuvant Chemotherapy

INTERVENTIONS:
Radiation: Preoperative SBRT for the Primary Lesion of Breast Cancer — SBRT for Primary Lesion of Breast Cancer, Radiation Dose: Primary Lesion ≤3 cm, GTV 24Gy/3F; Primary Lesion >3 cm, GTV 30Gy/5F.
  Arms: Neoadjuvant Chemoradiotherapy Group

SUMMARY:
This study focuses on preoperative treatment modalities for luminal-type locally advanced breast cancer. Based on modern precision radiotherapy technologies such as MRI-Linac, CyberKnife, and VMAT, it aims to compare the pCR rate, breast conserving surgery (BCS) rate, progression-free survival (PFS), and treatment-related side effects between preoperative neoadjuvant chemotherapy and preoperative neoadjuvant SBRT combined with chemotherapy in patients with this type of breast cancer. The goal is to provide new strategic options for the preoperative treatment of luminal-type locally advanced breast cancer.

DETAILED DESCRIPTION:
Breast cancer is a tumor with high tumor heterogeneity, and treatment outcomes vary significantly across different molecular subtypes. In recent years, the emergence of novel treatment methods has significantly improved the overall survival and progression-free survival of patients with early-stage, especially metastatic tumors. However, a portion of patients with locally advanced breast cancer (LABC) still have poor prognoses. As early as the 1970s, preoperative radiotherapy was applied to locally advanced breast cancer to increase resectability, but due to limitations in radiotherapy techniques and other factors, preoperative radiotherapy increased the incidence of acute toxic reactions and postoperative complications. Compared to traditional postoperative radiotherapy, neoadjuvant radiotherapy has several theoretical advantages, such as more precise tumor target localization, optimization of breast reconstruction radiotherapy strategies, increased tumor downstaging to improve breast-conserving surgery opportunities, and improved pathological complete response rates, potentially eliminating the need for breast surgery. With the advent of the era of precision radiotherapy, modern radiotherapy technologies have provided solutions to reduce the acute toxic reactions associated with preoperative radiotherapy. This study focuses on preoperative treatment modalities for luminal-type locally advanced breast cancer. It aims to compare the pCR rate, breast-conserving surgery (BCS) rate, progression-free survival (PFS), and treatment-related side effects between preoperative neoadjuvant chemotherapy and preoperative neoadjuvant SBRT combined with chemotherapy in these patients. The goal is to provide new strategic options for the preoperative treatment of luminal-type locally advanced breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically confirmed invasive breast cancer ;
2. Breast MRI showing stages IIB to IIIC (2017 AJCC 8th edition staging);
3. Clinical staging confirmed by chest MRI and/or axillary ultrasound, as well as CT scans of the neck, abdomen, and pelvis, and bone scintigraphy, including T and N staging and assessment of distant metastasis;
4. Karnofsky performance score ≥80 or ECOG performance status of 0-1;
5. No history of allergies to doxorubicin, cyclophosphamide, paclitaxel/docetaxel;
6. No prior exposure to radiotherapy, chemotherapy, endocrine therapy, targeted therapy, or immunotherapy.

Exclusion Criteria:

1. History of malignancy at other sites, excluding curable non-melanoma skin cancer and carcinoma in situ of the cervix;
2. Inability to complete MRI;
3. Inflammatory breast cancer;
4. Bilateral or multifocal primary tumors;
5. Active infection currently present; clinically evident heart disease; myocardial infarction or cerebrovascular accident within 6 months prior to enrollment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Estimated)
Dates: Start 2024-11-18 (Estimated); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
pCR | From enrollment to one month after surgery
  Pathological Complete Response Following Surgery

SECONDARY OUTCOMES:
Breast Conserving Surgery Rate | From enrollment to the completion of surgery
  Comparison of Breast Conserving Surgery Rates Between the Neoadjuvant Chemotherapy and Neoadjuvant Chemoradiotherapy Groups
PFS | From enrollment to the completion of the 3-year follow-up period
  Comparison of 3-Year Progression-Free Survival (PFS) Between the Neoadjuvant Chemotherapy and Neoadjuvant Chemoradiotherapy Groups
Adverse Event Incidence Rate | From enrollment to the completion of the 3-year follow-up period
  Comparison of Adverse Event Incidence Rates Between the Neoadjuvant Chemotherapy and Neoadjuvant Chemoradiotherapy Groups

CONTACTS AND LOCATIONS:
Overall Officials: Qian Peng, Phd, Principal Investigator — Sichuan Cancer Hospital and Research Institute; Junjie Li, Phd, Principal Investigator — Sichuan Cancer Hospital and Research Institute
Locations (1):
- Sichuan Cancer Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Vasmel JE, Charaghvandi RK, Houweling AC, Philippens MEP, van Asselen B, Vreuls CPH, van Diest PJ, van Leeuwen AMG, van Gorp J, Witkamp AJ, Koelemij R, Doeksen A, Sier MF, van Dalen T, van der Wall E, van Dam I, Veldhuis WB, Kirby AM, Verkooijen HM, van den Bongard HJGD. Tumor Response After Neoadjuvant Magnetic Resonance Guided Single Ablative Dose Partial Breast Irradiation. Int J Radiat Oncol Biol Phys. 2020 Mar 15;106(4):821-829. doi: 10.1016/j.ijrobp.2019.11.406. Epub 2019 Dec 5. PMID 31812720
- [Background] Nichols E, Kesmodel SB, Bellavance E, Drogula C, Tkaczuk K, Cohen RJ, Citron W, Morgan M, Staats P, Feigenberg S, Regine WF. Preoperative Accelerated Partial Breast Irradiation for Early-Stage Breast Cancer: Preliminary Results of a Prospective, Phase 2 Trial. Int J Radiat Oncol Biol Phys. 2017 Mar 15;97(4):747-753. doi: 10.1016/j.ijrobp.2016.11.030. Epub 2016 Nov 27. PMID 28244410
- [Background] Semiglazov VF, Topuzov EE, Bavli JL, Moiseyenko VM, Ivanova OA, Seleznev IK, Orlov AA, Barash NY, Golubeva OM, Chepic OF. Primary (neoadjuvant) chemotherapy and radiotherapy compared with primary radiotherapy alone in stage IIb-IIIa breast cancer. Ann Oncol. 1994 Sep;5(7):591-5. doi: 10.1093/oxfordjournals.annonc.a058929. PMID 7993833
- [Background] Ishitobi M, Suzuki O, Komoike Y, Ohsumi S, Nakahara S, Yagi T, Yoshinami T, Tomita Y, Inaji H. Phase II study of neoadjuvant anastrozole and concurrent radiotherapy for postmenopausal breast cancer patients. Breast Cancer. 2014 Sep;21(5):550-6. doi: 10.1007/s12282-012-0426-2. Epub 2012 Nov 2. PMID 23117619
- [Background] Bollet MA, Kirova YM, Antoni G, Pierga JY, Sigal-Zafrani B, Laki F, Campana F, Dendale R, Salmon R, Cottu P, Fourquet A. Responses to concurrent radiotherapy and hormone-therapy and outcome for large breast cancers in post-menopausal women. Radiother Oncol. 2007 Dec;85(3):336-45. doi: 10.1016/j.radonc.2007.10.003. Epub 2007 Oct 29. PMID 17967495
- [Background] Spring LM, Gupta A, Reynolds KL, Gadd MA, Ellisen LW, Isakoff SJ, Moy B, Bardia A. Neoadjuvant Endocrine Therapy for Estrogen Receptor-Positive Breast Cancer: A Systematic Review and Meta-analysis. JAMA Oncol. 2016 Nov 1;2(11):1477-1486. doi: 10.1001/jamaoncol.2016.1897. PMID 27367583
- [Background] Brackstone M, Palma D, Tuck AB, Scott L, Potvin K, Vandenberg T, Perera F, D'Souza D, Taves D, Kornecki A, Muscedere G, Chambers AF. Concurrent Neoadjuvant Chemotherapy and Radiation Therapy in Locally Advanced Breast Cancer. Int J Radiat Oncol Biol Phys. 2017 Nov 15;99(4):769-776. doi: 10.1016/j.ijrobp.2017.06.005. Epub 2017 Jun 20. PMID 28870785
- [Background] Roth SL, Audretsch W, Bojar H, Lang I, Willers R, Budach W. Retrospective study of neoadjuvant versus adjuvant radiochemotherapy in locally advanced noninflammatory breast cancer : survival advantage in cT2 category by neoadjuvant radiochemotherapy. Strahlenther Onkol. 2010 Jun;186(6):299-306. doi: 10.1007/s00066-010-2143-0. Epub 2010 May 21. PMID 20495968
- [Background] Riet FG, Fayard F, Arriagada R, Santos MA, Bourgier C, Ferchiou M, Heymann S, Delaloge S, Mazouni C, Dunant A, Rivera S. Preoperative radiotherapy in breast cancer patients: 32 years of follow-up. Eur J Cancer. 2017 May;76:45-51. doi: 10.1016/j.ejca.2017.01.022. Epub 2017 Mar 6. PMID 28267657
- [Background] Kim HJ, Noh WC, Lee ES, Jung YS, Kim LS, Han W, Nam SJ, Gong G-, Kim HJ, Ahn SH. Efficacy of neoadjuvant endocrine therapy compared with neoadjuvant chemotherapy in pre-menopausal patients with oestrogen receptor-positive and HER2-negative, lymph node-positive breast cancer. Breast Cancer Res. 2020 May 27;22(1):54. doi: 10.1186/s13058-020-01288-5. PMID 32460816
- [Background] Cataliotti L, Buzdar AU, Noguchi S, Bines J, Takatsuka Y, Petrakova K, Dube P, de Oliveira CT. Comparison of anastrozole versus tamoxifen as preoperative therapy in postmenopausal women with hormone receptor-positive breast cancer: the Pre-Operative "Arimidex" Compared to Tamoxifen (PROACT) trial. Cancer. 2006 May 15;106(10):2095-103. doi: 10.1002/cncr.21872. PMID 16598749
- [Background] Chow LWC, Morita S, Chow CYC, Ng WK, Toi M. Neoadjuvant palbociclib on ER+ breast cancer (N007): clinical response and EndoPredict's value. Endocr Relat Cancer. 2018 Feb;25(2):123-130. doi: 10.1530/ERC-17-0396. Epub 2017 Nov 20. PMID 29158285
- [Background] Alba E, Calvo L, Albanell J, De la Haba JR, Arcusa Lanza A, Chacon JI, Sanchez-Rovira P, Plazaola A, Lopez Garcia-Asenjo JA, Bermejo B, Carrasco E, Lluch A; GEICAM. Chemotherapy (CT) and hormonotherapy (HT) as neoadjuvant treatment in luminal breast cancer patients: results from the GEICAM/2006-03, a multicenter, randomized, phase-II study. Ann Oncol. 2012 Dec;23(12):3069-3074. doi: 10.1093/annonc/mds132. Epub 2012 Jun 6. PMID 22674146
- [Background] Cardoso F, Kyriakides S, Ohno S, Penault-Llorca F, Poortmans P, Rubio IT, Zackrisson S, Senkus E; ESMO Guidelines Committee. Electronic address: clinicalguidelines@esmo.org. Early breast cancer: ESMO Clinical Practice Guidelines for diagnosis, treatment and follow-updagger. Ann Oncol. 2019 Aug 1;30(8):1194-1220. doi: 10.1093/annonc/mdz173. No abstract available. PMID 31161190
- [Background] Gianni L, Pienkowski T, Im YH, Roman L, Tseng LM, Liu MC, Lluch A, Staroslawska E, de la Haba-Rodriguez J, Im SA, Pedrini JL, Poirier B, Morandi P, Semiglazov V, Srimuninnimit V, Bianchi G, Szado T, Ratnayake J, Ross G, Valagussa P. Efficacy and safety of neoadjuvant pertuzumab and trastuzumab in women with locally advanced, inflammatory, or early HER2-positive breast cancer (NeoSphere): a randomised multicentre, open-label, phase 2 trial. Lancet Oncol. 2012 Jan;13(1):25-32. doi: 10.1016/S1470-2045(11)70336-9. Epub 2011 Dec 6. PMID 22153890
- [Background] Alvarado-Miranda A, Arrieta O, Gamboa-Vignolle C, Saavedra-Perez D, Morales-Barrera R, Bargallo-Rocha E, Zinser-Sierra J, Perez-Sanchez V, Ramirez-Ugalde T, Lara-Medina F. Concurrent chemo-radiotherapy following neoadjuvant chemotherapy in locally advanced breast cancer. Radiat Oncol. 2009 Jul 11;4:24. doi: 10.1186/1748-717X-4-24. PMID 19591689
- [Background] Cortazar P, Zhang L, Untch M, Mehta K, Costantino JP, Wolmark N, Bonnefoi H, Cameron D, Gianni L, Valagussa P, Swain SM, Prowell T, Loibl S, Wickerham DL, Bogaerts J, Baselga J, Perou C, Blumenthal G, Blohmer J, Mamounas EP, Bergh J, Semiglazov V, Justice R, Eidtmann H, Paik S, Piccart M, Sridhara R, Fasching PA, Slaets L, Tang S, Gerber B, Geyer CE Jr, Pazdur R, Ditsch N, Rastogi P, Eiermann W, von Minckwitz G. Pathological complete response and long-term clinical benefit in breast cancer: the CTNeoBC pooled analysis. Lancet. 2014 Jul 12;384(9938):164-72. doi: 10.1016/S0140-6736(13)62422-8. Epub 2014 Feb 14. PMID 24529560
- [Background] Gradishar WJ, Moran MS, Abraham J, Abramson V, Aft R, Agnese D, Allison KH, Anderson B, Burstein HJ, Chew H, Dang C, Elias AD, Giordano SH, Goetz MP, Goldstein LJ, Hurvitz SA, Jankowitz RC, Javid SH, Krishnamurthy J, Leitch AM, Lyons J, Mortimer J, Patel SA, Pierce LJ, Rosenberger LH, Rugo HS, Schneider B, Smith ML, Soliman H, Stringer-Reasor EM, Telli ML, Wei M, Wisinski KB, Young JS, Yeung K, Dwyer MA, Kumar R. NCCN Guidelines(R) Insights: Breast Cancer, Version 4.2023. J Natl Compr Canc Netw. 2023 Jun;21(6):594-608. doi: 10.6004/jnccn.2023.0031. PMID 37308117
- [Background] Kuerer HM, Newman LA, Smith TL, Ames FC, Hunt KK, Dhingra K, Theriault RL, Singh G, Binkley SM, Sneige N, Buchholz TA, Ross MI, McNeese MD, Buzdar AU, Hortobagyi GN, Singletary SE. Clinical course of breast cancer patients with complete pathologic primary tumor and axillary lymph node response to doxorubicin-based neoadjuvant chemotherapy. J Clin Oncol. 1999 Feb;17(2):460-9. doi: 10.1200/JCO.1999.17.2.460. PMID 10080586
- [Background] Board, P.D.Q.A.T.E., Breast Cancer Treatment (PDQ®): Health Professional Version, in PDQ Cancer Information Summaries. 2002, National Cancer Institute (US): Bethesda (MD).
- [Background] Aldrich J, Canning M, Bhave M. Monitoring of Triple Negative Breast Cancer After Neoadjuvant Chemotherapy. Clin Breast Cancer. 2023 Dec;23(8):832-834. doi: 10.1016/j.clbc.2023.08.001. Epub 2023 Aug 5. PMID 37596146
- [Background] Nabieva N, Altmann F, Apel K, Baerens DT, Beha M, Belau A, Busch S, Guth D, Heinrich G, Kreiss-Sender J, Markmann S, Olbermann A, Oskay-Ozcelik G, Schuback B, Steinfeld-Birg D, Quiering C, Kiss F, Kreuzeder J, Nuti P, Schilling J. The Endocrine Treatment Landscape for Patients with HR+ HER2- Early-stage Breast Cancer in Germany Before the Introduction of CDK4/6 Inhibitor Therapy - A Real-World Analysis. Geburtshilfe Frauenheilkd. 2023 Jul 18;83(9):1127-1137. doi: 10.1055/a-2100-0643. eCollection 2023 Sep. PMID 37942358